CLINICAL TRIAL: NCT01573286
Title: Phase 1-2 Trial of Glucagon-like Peptide 2 (GLP-2) in Infants and Children With Intestinal Failure
Brief Title: Safety and Dosing Study of Glucagon-like Peptide 2 (GLP-2) in Infants and Children With Intestinal Failure
Acronym: GLP-2-01
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: GLP-2 Drug product stability concerns
Sponsor: Alberta Children's Hospital (Other)
Collaborators: Stollery Children's Hospital (Other); The Hospital for Sick Children (Other); British Columbia Children's Hospital (Other)
Responsible Party: Principal Investigator, David Sigalet MD PhD, Adjunct Professor, Division of Pediatric Surgery, Alberta Children's Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GLP-2-01; 150979 (Other: Health Canada)
Record Dates: First submitted 2012-04-05; First posted 2012-04-09 (Estimated); Last update posted 2014-12-23 (Estimated); Status verified 2014-12

CONDITIONS: Intestinal Failure; Short Bowel Syndrome
Keywords: Infant Nutrition Disorders; Childhood nutrition disorders; malnutrition; post surgical syndromes; necrotising enterocolitis; intestinal atresia; gastroschisis
MeSH Terms: conditions — Intestinal Failure; Short Bowel Syndrome; Infant Nutrition Disorders; Malnutrition; Enterocolitis, Necrotizing; Intestinal Atresia; Gastroschisis | interventions — Glucagon-Like Peptide 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intestinal Failure in children (>1 year) (Experimental): Children requiring parenteral nutrition for >30% of calories more than 1 year (365) days post surgery will be eligible for treatment with Glucagon-like peptide 2 (20 ug/kg/day) for 6 weeks
  Interventions: Drug: Glucagon-Like Peptide 2
- GLP-2 in Infants (<1 year of age) (Experimental): Infants under one year of age with congenital anomalies, or intestinal resection, leaving them with anatomic short bowel syndrome (total remaining small intestine less than 40 % of predicted for gestational age) or with intestinal resection or repaired gastroschisis who have demonstrated dependence on parenteral nutrition at 45 days post operation with the requirement for >50% of calories by PN (independent of the length of remnant small intestine) will be eligible for treatment with Glucagon-like peptide 2, at a dose of 5, 10 or 20 ug/kg/day.
  Interventions: Drug: Glucagon like peptide-2

INTERVENTIONS:
Drug: Glucagon-Like Peptide 2 — Patients will be treated with 20 ug/kg/day GLP-2, in two doses, given subcutaneously for 3 days (Phase 1). If the treatment is well tolerated, GLP-2 will be continued for a total of 42 days.
  Other Names: Glucagon-like peptide-2 (Lot: IC-115) Mfg. University of Calgary
  Arms: Intestinal Failure in children (>1 year)
Drug: Glucagon like peptide-2 — Patients will treated with 5, 10 or 20 ug/kg/day of GLP-2, given twice daily by subcutaneous injection. The initial cohort of patients will be treated at 5 ug/kg (n=6), and if this dose is seen to be safe, and levels appropriate, the next group of 6 will be treated at 10 ug/kg/day. If this dose is seen to be safe, and levels appropriate, the final group of 6 will be treated at 20 ug/kg/day.
  Patients will be given GLP-2 at the assigned dose, subcutaneously for 3 days (Phase 1). If the treatment is well tolerated, GLP-2 will be continued, at the same dose, for a total of 42 days.
  Other Names: Glucagon-like peptide-2 (Lot: IC-115) Mfg. University of Calgary
  Arms: GLP-2 in Infants (<1 year of age)

SUMMARY:
This protocol outlines a randomized,open label trial examining the safety, pharmacology and efficacy of Glucagon like peptide 2 (GLP-2) in infants and children with intestinal failure. The investigators hypothesize that GLP-2 given subcutaneously in these patients will be well tolerated, and have similar metabolism to what has been shown in adults. The investigators also expect to show an improvement in the tolerance of enteral nutrition, and a decreased requirement for intravenous feeding.

DETAILED DESCRIPTION:
GLP-2 (1-33) is a naturally occurring peptide which is important in controlling the function of the intestine. In previous studies our group has shown that serum levels of GLP-2 correlate with intestinal function in human neonates. Low levels of GLP-2 are predictive of intestinal malabsorption and the development of the so called "Short Bowel Syndrome". GLP-2 has been shown to be specifically trophic for the GI tract, especially for the small intestine.

This proposal outlines a Phase 1 and 2 trial using subcutaneous administration, twice daily of GLP-2 in human infants and children with Intestinal Failure, typically from Short Bowel Syndrome, using varying doses, assigned in a prospective, randomized protocol, with open label monitoring.

The investigational plan is to begin with the Phase 1 trial, administering GLP 2 at varying doses (infants assigned to doses of 5,10, or 20 μg/kg/day, children greater than 1 year dosed at 20 μg/kg/day, given via twice daily subcutaneous injection).

Eligible subjects will be infants (less than 12 months corrected gestational age) with either major resection (remaining small intestine less than 40% of predicted length for gestational age), or demonstrated intestinal failure after intestinal resection/abdominal surgery/gastroschisis (Requirement for parenteral nutrition greater than 50% of total calories, more than 45 days after the last surgery).

Infants will be allocated sequentially to a group (n = 6 per group) treated with GLP-2 at 5,10, or 20 μg/kg/day.

Older children (greater than 1 year of age), requiring PN for >30% calories> one year post surgery will also be eligible; these patients will be dosed at 20 μg/kg/day (via twice daily subcutaneous injection) n= 7.

Patients will be followed on the principle of intention to treat after initial randomization. The endpoints will be monitoring for safety, and recording of adverse events and a pharmacokinetic profile at 3 days.

If the hormone is well tolerated these studies will be extended into a phase 2 study, for an additional 39 days; monitoring safety, patient tolerance of enteral nutrition, growth, citrulline levels, nutrient absorptive capacity, liver function and repeat pharmacokinetic studies.

ELIGIBILITY:
Inclusion Criteria:

* Infants (< 1 year corrected gestational age) Infants with congenital anomalies, or intestinal resection, leaving them with anatomic short bowel syndrome (total remaining small intestine less than 40 % of predicted for gestational age) will be eligible for treatment in the immediate post-operative period.
* Infants with intestinal resection or repaired gastroschisis who have demonstrated dependence on parenteral nutrition at 45 days post operation with the requirement for >50% of calories by PN (independent of the length of remnant small intestine).
* Children (> 1 year corrected gestational age) Children with a requirement for >30% of calories by PN more than 1 year (365) days post surgery will be eligible.

Exclusion Criteria:

* Significant extra-intestinal disease (e.g., grade IV intraventricular hemorrhage, severe hypoxic encephalopathy);
* Significant cardiovascular, hemodynamic or respiratory instability, as noted by 1) the requirement for dopamine > 4 mcg/kg/min, 2) high frequency ventilatory support, 3) extracorporeal membrane oxygenation.
* Hepatic disease defined as direct bilirubin > 100 umol/L (5.2 mg/dL)
* Renal disease defined as BUN > 80 or creatinine > 90 μmol/L (1.5 mg/dL)
* Inborn errors of metabolism necessitating protein restriction or other special diet;
* Ongoing sepsis syndrome, as noted by refractory hypotension, thrombocytopenia, acidosis, and/or bacteremia.
* Primary motility defect such as intestinal pseudo-obstruction.
* Absorptive defects (such as microvillus inclusion disease)
* Females who are post-pubertal must agree to comply with measures to prevent pregnancy during the study phase.
* Coagulopathy which precludes the use of subcutaneous injections.
* Allergy to GLP-2 or any of the constituent of the GLP-2 IC-115 preparation.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 13 (Actual)
Dates: Start 2012-01; Primary Completion 2014-08 (Actual); Study Completion 2015-08 (Estimated)

PRIMARY OUTCOMES:
Frequency of Adverse events | One year
  During active drug administration, patients will be monitored daily for serious adverse events. Patients will also be monitored (daily, if inpatients, bi weekly if outpatients) for clinically significant changes in safety data, vital signs, physical examination,and injection site reactions. Laboratory values of liver function and renal function will be monitored weekly for inpatients and bi weekly for outpatients.
  Following discontinuation of the treatment, patients will be monitored at 1 ,6 and 12 months post completion of the therapy.
Pharmacokinetics (Peak serum level. Area under the curve | Done on Day 3 and 42
  On days 3 and 42 of the trial, GLP-2 levels will be drawn at time 0 (before injection), 45,90 and 180 minutes post injection. Results will be analyzed for peak levels, and AUC.

SECONDARY OUTCOMES:
Changes in the Enteral Caloric intake | one year
  During active drug administration, changes in the proportion of total enteral calories tolerated (Including discontinuation of parenteral nutrition) will be monitored twice weekly (hospital inpatients) and weekly (for outpatients). Following the phase of active treatment, patients will be followed at 1, 6, and 12 months.
Nutritional Parameters | one year
  During the phase of active treatment, nutritional parameters; weight gain, maintenance of growth (z scores), Liver function, albumin, protein levels, C-reactive protein, electrolytes, renal function (creatinine levels) will be monitored twice weekly (hospital inpatients) and weekly (for outpatients). Following the phase of active treatment, patients will be followed at 1, 6, and 12 months.
Mucosal Morphology | 6 weeks
  If procedures requiring sedation or surgery are done during the phase of active drug administration, intestinal biopsies will be requested, to quantify changes in crypt cell proliferation and apoptosis index, and intestinal morphology (villus height and/or crypt depth) between pre-treatment surgical samples, and specimens obtained while under treatment.
Intrinsic GLP-2 Production | One year
  At the beginning of the active treatment, and during week 5, intrinsic meal stimulated GLP-2 production will be assessed. During followup, these values will be assessed at 1,6 and 12 months post-treatment
Septic Episodes | 6 weeks
  During the treatment phase, the number of septic episodes, and the type of infecting organisms will be recorded.
Serum Citrulline Levels | One year.
  Citrulline levels as a measure of intestinal mucosal mass will be assessed at time 0, and on the last day of active treatment. During followup, these values will be assessed at 1,6 and 12 months post-treatment

CONTACTS AND LOCATIONS:
Overall Officials: David Sigalet, MD PhD, Study Director — Alberta Children's Hospital
Locations (4):
- Canada (4):
  - Alberta Children's Hospital, Calgary, Alberta
  - Stollery Children's Hospital, Edmonton, Alberta
  - British Columbia Children's Hospital, Vancouver, British Columbia
  - Hospital for Sick Children, Toronto, Ontario

REFERENCES:
- [Background] Sigalet DL, de Heuvel E, Wallace L, Bulloch E, Turner J, Wales PW, Nation P, Wizzard PR, Hartmann B, Assad M, Holst JJ. Effects of chronic glucagon-like peptide-2 therapy during weaning in neonatal pigs. Regul Pept. 2014 Jan 10;188:70-80. doi: 10.1016/j.regpep.2013.12.006. Epub 2013 Dec 22. PMID 24368164
- [Result] Sigalet DL, Lam V, Karnik V, Brindle M, Boctor D, Casey LW, Dicken B, Butterworth S, Stoffman S,de Heuval E, Wright-wilson G, Wallace L. Safety and Dosing Study of Glucagon-like Peptide 2 (GLP-2) in Children With Intestinal Failure DDW Abstract presented at DDW 2014, Chicago IL